### INFORMED CONSENT FORM

# **I-Providing Information About Research**

A responsible researcher, Istanbul University School of Dentistry Oral & Maxillofacial radiology, faculty member Prof. Dr. Ilknur Özcan Department of this study; 442 26/09/2019 date and with the approval of the Ethics Committee, Dt. A. is carried out by Faruk Ertürk.

- Our Valued Volunteer
- This study Temporomandibular Dysfunction (TMJ Diseases) in the treatment of diseases of low-dose laser treatment was to investigate the effectiveness of the method.
- The topics that comprise the content of the study are presented below.
- 1. Demographic Information
- (In the study, no personal information is not requested.)
- 2. Disease-Related Assessments
- 3. Made For Viewing Values For Transform
- The application lasts more than 15 minutes.
- Principal investigator and contact information

Dr. Ilknur ÖZCAN - Istanbul University Faculty of dentistry, department of oral and maxillofacial radiology – iozcan@istanbul.edu.tr - 0212 414 20 20

Other Researchers

Dr. bilge GÖKÇEN ROHLIG - Istanbul University, Faculty of dentistry, department of Prosthodontics

LEC. See. Dr. Hülya black-headed Goshawk - Istanbul University Faculty of dentistry, department of oral and maxillofacial radiology

Dt. A. Faruk ERTURK - Istanbul University Faculty of dentistry, department of oral and maxillofacial radiology

# PLEASE, READ CAREFULLY!

You have been invited to participate in a clinical study for purposes of scientific research. Before you agree to take part in this study done what is the purpose of the study were fully informed about the research and wants to be your decision after you fully understand that you are required to give freely. This disclosure form in question in order to introduce the research in detail and tailored to you. Please read this form carefully. You are free not to participate in this research project. Participation in the study is voluntary. To participate in the survey if you agree, by signing the form, your operations can continue.

NAME OF RESEARCH

Temporomandibular Dysfunction (Jaw Bone Disease) In Patients With Different Treatment Techniques For Myofascial Trigger Points (Excessive Masticatory Muscles Twitch Points) Of The Impact Of Prospective (Forward-Looking) Examination

# NUMBER OF VOLUNTEERS

This research is projected to take place in the total number of stop 60.

### DURATION OF PARTICIPATION IN THE RESEARCH

To take part in this research, the prescribed period is 24 months.

# PURPOSE OF THE STUDY

In this study, TMD and occlusal splints in the treatment of low-dose laser therapy (lll) the use of, as a result of USG at certain intervals and other parameters by evaluating changes in the chewing muscles, which is the treatment method is more efficient and at the same time also evaluating the parameter which is the parameters that are used in its own right because it demonstrates that scientific resources is intended to contribute to is more effective.

# RESEARCH METHOD

To all the volunteers that will participate in the research pre-treatment of the joint examination and Ultrasonographic examination (USG) shall be governed by. The USG open and closed mouth in the application, the measurements made will be deducted from the note intervals of the left and right joints. At the same time the right and left masseter (masticatory muscle) and tight closing in closing free Nov thicknesses measured separately for all groups and will be deducted from the note.

To participate in the research volunteers will be divided into 2 groups(Laser Group: I.; Splint Group: II. Group). A group of 30 people randomly selected low-dose Laser be applied again to 30 will be chosen at random II. the group and the group prepared by the conventional method will be applied to record the night. After treatment 1.month 3.months and 6.month for checkups and examination data obtained by applying joint tests are invoked by patients for control purposes the Note will be deducted from the USG. Laser splint after the investigation and the findings compared with each other groups, low-dose efficacy of laser therapy will be analyzed statistically.

### TREATMENTS TO BE APPLIED IN THE RESEARCH

Research record at night and laser therapy will be applied.

### THE POTENTIAL BENEFITS FROM THE RESEARCH

Treatment method in the treatment of TMD, which is more efficient and can be assessed more accurately by the parameters of what they are putting forward the success of the treatment in patients with TMD.

# EXPECTED FROM THE RESEARCH, POTENTIAL RISKS/LOSSES

Applications and LLL night guard, non-invasive (non-invasive) is a process and can be applied safely even for pregnant women. So the methods that will be used in research does not pose any risk.

# II-the rights of the volunteer to be given information about

### COVERING THE EXPENSES AND PAYMENTS

For expenses that may result from this research or to participate in the research, no fee shall be required of you.

# INSTITUTIONS THAT SUPPORT RESEARCH

Institutions that support research, Istanbul University scientific research projects (BAP)is.

### VOLUNTEERS, WHETHER ANY PAYMENT

Will not provide any financial contribution you or your legal representatives.

# CONFIDENTIALITY OF INFORMATION

Information about you obtained during the research period, which for you with a special code number will be saved. You will not be asked from you, no personal information(ID number, etc.) the results of the research will be used only for scientific purposes. Research credentials will not be given even aired. However, polling the audience of those who do the necessary research, ethical committees and authorities will be able to access your personal information. When you want your own information, you will be able to reach after the analysis of the data.

### VOLUNTEER RESPONSIBILITIES AND CONDITIONS TO BE LEFT OUT OF THE RESEARCH

If you provide incorrect information intentionally, we aksatman research program, the researcher can get out of your research without your permission. However, the research is also left out of about you, your identity remain confidential medical data for scientific purposes in a way that may be of use.

# REFUSE TO PARTICIPATE IN RESEARCH OR LEAVE THE STATUS

Taking part in this research is entirely voluntary. You may leave the study or refuse to take part in the research at any stage; you can give up or you refuse to take part in the study after you join, you may use for scientific purposes in a way that your identity remain confidential medical data.

### Volunteers Statement

Mr D. t Faruk ERTÜRK A. by Istanbul University Faculty of Dentistry Oral and maxillofacial radiology, department of medical research made a research related to this by stating that the above information will be transferred to me. This information is then to study such a "voluntary", as I was invited. If I'm involved in this research project the physician should remain with the confidentiality of the information that belongs to me during this research can be approached with great care and respect I believe. The results of the research for educational and scientific purposes during the use of my personal information will be protected with the necessary care it was given enough confidence to me about.

I can withdraw from the research without showing any reason during the execution of the project. (However, researchers from the research fall on the sword to leave a difficult situation and I'm aware that I would be appropriate prior to reporting) is also the condition that my medical condition is not in any harm by the researcher out of the research, too, I can.

For research to be made on the expenditure side, I am not getting any monetary responsibility. Me a payment will be made.

Either directly or indirectly, arising from the application of research I develop any health problems that may occur if the necessary assurance was given that any medical intervention will be provided. (This is under load I'm not getting medical treatment in connection with a monetary).

When faced with a health problem during the investigation; at any time, Dt. To A. Faruk Ertürk, oral and maxillofacial radiology Faculty of Dentistry and IU the name of-0505 782 88 44I know that I can call from. I may not agree and I don't have to participate in this research project. I'm not encountering a compelling research about joining behavior. If I refuse to participate if the physician of this condition will not bring any harm to my relationship with medical care and I know that.

To me all comments are understood in detail. On my own thinking in this research project mentioned at the end of a certain period of "voluntary" as I took the decision to take part. The invitation with great satisfaction in volunteering on this subject and I agree.

A paper copy of the signed form will be given to me.

### **VOLUNTARY CONSENT FORM**

The volunteer survey that indicates the information above must be given before I read the text. Written and oral comments made to me about them. Under these conditions, no pressure on my own volition without coercion to participate in a clinical research question and I agree.

Volunteer Name-Last Name/ Signature/Date/ address (if available phone no. no fax,...)

The research team located and a competent researcher

Name-Last Name/ Signature/ Date

Becomes the name of the person who witnessed the process if necessary-Your Last Name/Signature/Date/ address (if available phone no. no fax,...)

If necessary, the legal representative's Name-Last Name/ Signature/Date/ address (if available phone no. no fax,...)